CLINICAL TRIAL: NCT01634269
Title: Medtronic MDT-2111 CoreValve Japan 23mm Study
Brief Title: Clinical Evaluation of MDT-2111 in Subjects With Small Aortic Annuli and Symptomatic Severe Aortic Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT-2111 23 mm trial
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Aortic Valve Stenosis
Keywords: Valvular Heart Disease; Severe Aortic Stenosis; Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MDT-2111 TAVI 23 mm (Experimental): Subjects with small annuli and symptomatic severe AS deemed difficult for surgical intervention.
  Interventions: Device: MDT-2111 TAVI 23 mm

INTERVENTIONS:
Device: MDT-2111 TAVI 23 mm — Device: 23 mm MDT-2111 System for Transcatheter Aortic Valve Implantation (TAVI) Transcatheter Aortic Valve Implantation (TAVI) using the 23 mm MDT-2111 system.

SUMMARY:
The primary objective of the present trial is to demonstrate the safety and effectiveness of the MDT-2111 in the treatment of symptomatic severe aortic stenosis in subjects with small aortic annuli and deemed difficult for surgical operation.

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate the effectiveness and safety of the MDT-2111 TAV system in subjects with small annuli and symptomatic severe AS deemed difficult for surgical intervention. The primary endpoint is a composite of functional effectiveness as measured by improvement of at least 1 New York Heart Association (NYHA) class from baseline to 6 months and anatomical effectiveness as measured by Effective Orifice Area (EOA) ≥1.0 cm² at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have co-morbidities such that one cardiologist and one cardiac surgeon agree that medical factors preclude operation, based on a conclusion that the probability of death or serious morbidity exceeds the probability of meaningful improvement.
2. Subject has senile degenerative aortic valve stenosis with:

   mean gradient > 40 mmHg or jet velocity greater than 4.0 m/s by either resting or dobutamine stress echocardiogram, or simultaneous pressure recordings at cardiac catheterization (either resting or dobutamine stress), AND an initial aortic valve area of ≤ 0.8 cm² (or aortic valve area index ≤ 0.5 cm²/m²) by resting echocardiogram.
3. Subject is symptomatic from his/her aortic valve stenosis, as demonstrated by NYHA Functional Class Class III or greater. If screening committee agrees the eligibility of a patient with class II , based on medical factors, he/she can be enrolled.
4. Patient has been informed of the nature of the trial and has signed an Informed Consent Form.
5. Patient agrees to comply with specified follow-up evaluations and to return to the same investigational site where the procedure was performed.

Exclusion Criteria:

1. Evidence of an acute myocardial infarction ≤ 30 days prior to the intended treatment.
2. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to the procedure.
3. Blood dyscrasias as defined:

   * Leukopenia (WBC count < 1,000 cells/mm³)
   * Thrombocytopenia (platelet count <50,000 cells/mm³)
   * History of bleeding diathesis or coagulopathy
   * Hypercoagulable states
4. Untreated clinically significant coronary artery disease requiring revascularization.
5. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support.
6. Need for emergency surgery for any reason.
7. Severe ventricular dysfunction with left ventricular ejection fraction (LVEF) < 20% as measured by resting echocardiogram.
8. Recent (within 6 months) cerebrovascular accident (CVA) or transient ischemic attack(TIA).
9. End stage renal disease requiring chronic dialysis.
10. GI bleeding within the past 3 months.
11. A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated:

    * Aspirin
    * Ticlopidine
    * Heparin
    * Contrast media
    * Nitinol (titanium and nickel alloy)
12. Ongoing sepsis, including active endocarditis.
13. Subject refuses a blood transfusion.
14. Life expectancy < 12 months due to associated non-cardiac co-morbid conditions.
15. Other medical, social, or psychological conditions that in the opinion of an Investigator precludes the subject from appropriate consent.
16. Severe dementia (resulting in either inability to provide informed consent for the trial/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits).
17. Currently participating in an investigational drug or another device trial. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
18. Symptomatic carotid or vertebral artery disease.
19. Native aortic annulus size < 18 mm or > 20 mm per the screening diagnostic imaging.
20. Pre-existing prosthetic heart valve in any position.
21. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation).
22. Mitral regurgitation (moderate to severe) or severe tricuspid regurgitation.
23. Moderate to severe mitral stenosis.
24. Hypertrophic obstructive cardiomyopathy.
25. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
26. Severe basal septal hypertrophy with an outflow gradient.
27. Ascending aorta diameter > 34 mm
28. Congenital bicuspid or unicuspid valve verified by echocardiography.
29. For patients with native coronary artery dependent circulation:

    * Sinus of valsalva width < 25 mm OR
    * Height of the left or right coronary sinus of valsalva (to the tubular aorta) < 15mm.
30. Femoral or iliac artery of the first choice corresponding to any one of the following:

    * Angle at aortic root (the angle between aortic valve annulus plane and horizontal plane/vertebra) exceeds 70°.
    * Vessel diameter of femoral or iliac artery is less than 6 mm.
    * Aorta has severe calcification, excess tortuosity or severe atherosclerosis.
    * Transarterial access not able to accommodate an 18Fr sheath.
31. Subclavian artery of the second choice corresponding to any one of the following:

    * Angle at aortic root (the angle between aortic valve annulus plane and horizontal plane/vertebra) exceeds 70° (in the case of left subclavian artery) and 30° (in the case of right subclavian artery).
    * Vessel diameter of subclavian artery is less than 6 mm.
    * Transarterial access not able to accommodate an 18Fr sheath.
32. Direct Aortic Artery as third line choice of access. Patients are excluded from Direct Aortic access if:

    * Access site is less than 6 cm from the aortic valve basal plane
    * Access site has calcification or porcelain aorta
    * Access site and delivery trajectory contain RIMA or patent RIMA graft

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2014-02 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshi Sawa, Professor, Principal Investigator — Osaka University Hospital
Locations (4):
- Japan (4):
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Saitama Medical University, Hidaka, Saitama

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sawa Y, Torikai K, Kobayashi J, Niinami H, Kuratani T, Maeda K, Kanzaki H, Komiyama N, Tanaka Y, Zhang A, Saito S. Midterm Outcomes With a Self-Expandable Transcatheter Heart Valve in Japanese Patients With Symptomatic Severe Aortic Stenosis. Circ J. 2017 Jul 25;81(8):1108-1115. doi: 10.1253/circj.CJ-17-0112. Epub 2017 Mar 17. PMID 28321003

RESULTS

PARTICIPANT FLOW:
Groups:
- MDT-2111 TAVI 23 mm: Transcatheter Aortic Valve Implantation (TAVI) using the 23 mm MDT-2111 system.
Period: Overall Study
Arm/Group | MDT-2111 TAVI 23 mm
Started | 20
30 Days | 20
6 Month | 20
12 Month | 20
24 Month | 18
Completed | 18
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | MDT-2111 TAVI 23 mm
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.0 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 1
Region of Enrollment [Number; unit: participants]
  Japan | 20
NYHA Class [Number; unit: participants] — NEW YORK HEART ASSOCIATION CLASSIFICATION (NYHA) Class I Subject with cardiac disease but without resulting limitations of physical activity. Class II Subjects with cardiac disease resulting in slight limitation of physical activity. Class III Subjects with cardiac disease resulting in marked limitation of physical activity. Class IV Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  participants
    NYHA Class II | 0
    NYHA Class III | 19
    NYHA IV | 1
STS Score [Mean (Standard Deviation); unit: percent] — The Society of Thoracic Surgeons (STS) risk model predicts the risk of operative mortality and morbidity after adult cardiac surgery on the basis of patient demographic and clinical variables. After information has been entered on a given case, the online STS risk calculator provides a risk percentage for each of the outcomes. The risk percentage estimates the chance of a specific outcome for a patient with the indicated risk factors. A higher score indicates a higher risk. A lower score indicates a lower risk.
  percent | 7.0 (3.3)
Logistic EuroScore [Mean (Standard Deviation); unit: percent] — The European System for Cardiac Operative Risk Evaluation (EuroSCORE) is a method of calculating predicted operative mortality for patients undergoing cardiac surgery. If a risk factor is present, a weight/number is assigned. The weights are added to give an approximate percent of predicted mortality. A higher score indicates a higher risk. A lower score indicates a lower risk.
  percent | 22.3 (10.1)
Body Surface Area [Mean (Standard Deviation); unit: m²] | 1.4 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Composite Score of Change in New York Heart Association (NYHA) Class and Effective Orifice Area (EOA).
Description: The primary endpoint is a composite of functional effectiveness as measured by improvement of at least 1 NYHA class from baseline to 6 months and anatomical effectiveness as measured by Effective Orifice Area (EOA) ≥1.0 cm² at 6 months.
Time Frame: baseline and 6 months
Population: Implanted subjects
Measure: Number; unit: percentage of participants analyzed
Groups:
- All Implanted Subjects: The Implanted population consisted of all As Treated Subjects who underwent an index procedure and were implanted with the MDT-2111 TAVI 23 mm device.
- Iliofemoral Implanted Subjects: The IF Implanted population consisted of all IF As Treated Subjects who underwent an index procedure and were implanted with the MDT-2111 device.
Arm/Group | All Implanted Subjects | Iliofemoral Implanted Subjects
Number analyzed (Participants) | 20 | 16
percentage of participants analyzed | 75.0 | 87.5
Statistical Analysis 1: Comparison: Iliofemoral Implanted Subjects; Test type: Superiority or Other; p = 0.002, Exact binomial; Proportion of IF implanted subjects = 87.5, 95.0% CI 2-sided [61.7 to 98.4]

2. Secondary Outcome: New York Heart Classification (NYHA) Over Time
Description: NEW YORK HEART ASSOCIATION CLASSIFICATION (NYHA) Class I: Subject with cardiac disease but without resulting limitations of physical activity.
  Class II: Subjects with cardiac disease resulting in slight limitation of physical activity.
  Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
Time Frame: 30 days
Population: All Implanted Subjects
Measure: Number; unit: percentage of participants analyzed
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
percentage of participants analyzed
  NYHA I | 45.0
  NYHA II | 50.0
  NYHA III | 5.0
  NYHA IV | 0.0
  Death | 0.0

3. Secondary Outcome: New York Heart Classification (NYHA) Over Time
Description: as for outcome 2
Time Frame: 6 months
Population: All Implanted Subjects
Measure: Number; unit: percentage of participants analyzed
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
percentage of participants analyzed
  NYHA I | 55.0
  NYHA II | 45.0
  NYHA III | 0.0
  NYHA IV | 0.0
  Death | 0.0

4. Secondary Outcome: New York Heart Classification (NYHA) Over Time
Description: as for outcome 2
Time Frame: 12 months
Population: All Implanted Subjects
Measure: Number; unit: percentage of participants analyzed
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
percentage of participants analyzed
  NYHA I | 40.0
  NYHA II | 60.0
  NYHA III | 0.0
  NYHA IV | 0.0
  Death | 0.0

5. Secondary Outcome: New York Heart Classification (NYHA) Over Time
Description: as for outcome 2
Time Frame: 24 months
Population: All Implanted Subjects
Measure: Number; unit: percentage of participants analyzed
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 19
percentage of participants analyzed
  NYHA I | 47.4
  NYHA II | 47.4
  NYHA III | 0.0
  NYHA IV | 0.0
  Death | 5.3

6. Secondary Outcome: Major Adverse Cardiovascular and Cerebrovascular Event (MACCE)
Description: MACCE is defined as a composite of:
  * all-cause death
  * myocardial infarction (MI)
  * all stroke, and
  * reintervention (defined as any cardiac surgery or percutaneous reintervention catheter procedure that repairs, otherwise alters or adjusts, or replaces a previously implanted valve)
Time Frame: 0 day to 30 days
Population: The Kaplan-Meier Method was used to calculate the number.
Measure: Number; unit: prob of freedom from event @ 30 days
Groups:
- As Treated Subjects: The As Treated (AT) population was defined as subjects with an attempted implant procedure, identified as subject entry to the procedure room and any of the following occurrences: anesthesia administered, vascular line placed, transesophageal echo (TEE) placed, or any monitoring line placed.
Arm/Group | As Treated Subjects
Number analyzed (Participants) | 20
prob of freedom from event @ 30 days | 100

7. Secondary Outcome: Major Adverse Cardiovascular and Cerebrovascular Event (MACCE)
Description: as for outcome 6
Time Frame: 0 day to 6 months
Population: The Kaplan-Meier Method was used to calculate the number.
Measure: Number; unit: prob of freedom from event @ 183 days
Arm/Group | As Treated Subjects
Number analyzed (Participants) | 20
prob of freedom from event @ 183 days | 95.0

8. Secondary Outcome: Major Adverse Cardiovascular and Cerebrovascular Event (MACCE)
Description: as for outcome 6
Time Frame: 0 day to 12 months
Population: The Kaplan-Meier Method was used to calculate the number.
Measure: Number; unit: prob of freedom from event @ 365 days
Arm/Group | As Treated Subjects
Number analyzed (Participants) | 20
prob of freedom from event @ 365 days | 95.0

9. Secondary Outcome: Major Adverse Cardiovascular and Cerebrovascular Event (MACCE)
Description: as for outcome 6
Time Frame: 0 day to 24 months
Population: The Kaplan-Meier Method was used to calculate the number.
Measure: Number; unit: prob of freedom from event @ 730 days
Arm/Group | As Treated Subjects
Number analyzed (Participants) | 20
prob of freedom from event @ 730 days | 90.0

10. Secondary Outcome: Device Success as Defined in the Description.
Description: The following components must be satisfied for device success:
  1. successful vascular access, delivery and deployment of device and successful retrieval of delivery system
  2. correct position of device in the proper anatomical location
  3. EOA≥1.0 cm² AND mean gradient <20 mmHg or peak velocity <3 m/s, without moderate or severe AR
  4. only one valve implanted.
Time Frame: after procedure or discharge
Population: This includes subjects with an index procedure. Index procedure is defined as the first procedure that Medtronic MDT-2111 TAV system delivery catheter is introduced.
Measure: Number; unit: percentage of participants analyzed
Groups:
- As Treated (AT) Subjects With Index Procedure: The (AT) population with Index Procedure was defined as subjects with an attempted implant procedure, identified as subject entry to the procedure room and any of the following occurrences: anesthesia administered, vascular line placed, transesophageal echo placed, or monitoring line placed. Index procedure was defined as introduction of the MDT-2111 TAV system delivery catheter.
Arm/Group | As Treated (AT) Subjects With Index Procedure
Number analyzed (Participants) | 20
percentage of participants analyzed | 65.0

11. Secondary Outcome: Procedural Success, Defined as Device Success and Absence of In-hospital MACCE
Description: Procedural success is defined as device success and absence of in-hospital MACCE.
Time Frame: from admission for procedure to discharge
Population: as for outcome 10
Measure: Number; unit: percent
Groups:
- As Treated Subjects With Index Procedure: The (AT) population with Index Procedure was defined as subjects with an attempted implant procedure, identified as subject entry to the procedure room and any of the following occurrences: anesthesia administered, vascular line placed, transesophageal echo placed, or monitoring line placed. Index procedure was defined as introduction of the MDT-2111 TAV system delivery catheter.
Arm/Group | As Treated Subjects With Index Procedure
Number analyzed (Participants) | 20
percent | 65.0

12. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Mean Gradient
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
mmHg | 16.8 (4.8)

13. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Mean Gradient
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
mmHg | 17.1 (7.7)

14. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Mean Gradient
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
mmHg | 15.2 (5.6)

15. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Mean Gradient
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 18
mmHg | 13.7 (5.6)

16. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Effective Orifice Area (EOA)
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
cm² | 1.2 (0.3)

17. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Effective Orifice Area (EOA)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
cm² | 1.2 (0.3)

18. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Effective Orifice Area (EOA)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 19
cm² | 1.2 (0.3)

19. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Effective Orifice Area (EOA)
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 16
cm² | 1.3 (0.3)

20. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Left Ventricular Ejection Fraction (LVEF)
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
percent | 64.5 (6.5)

21. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Left Ventricular Ejection Fraction (LVEF)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
percent | 66.8 (5.4)

22. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Left Ventricular Ejection Fraction (LVEF)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
percent | 67.5 (7.9)

23. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Left Ventricular Ejection Fraction (LVEF)
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 18
percent | 67.9 (4.9)

24. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Total Aortic Regurgitation (Transvalvular & Paravalvular) (Total AR)
Time Frame: 30 days
Measure: Number; unit: percentage of participants analyzed
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
percentage of participants analyzed
  None | 10.0
  Trace | 0.0
  Mild | 75.0
  Moderate | 15.0
  Severe | 0.0

25. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Total Aortic Regurgitation (Transvalvular & Paravalvular) (Total AR)
Time Frame: 6 months
Measure: Number; unit: percentage of participants analyzed
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
percentage of participants analyzed
  None | 0.0
  Trace | 30.0
  Mild | 55.0
  Moderate | 15.0
  Severe | 0.0

26. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Total Aortic Regurgitation (Transvalvular & Paravalvular) (Total AR)
Time Frame: 12 months
Measure: Number; unit: percentage of participants analyzed
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
percentage of participants analyzed
  None | 5.0
  Trace | 15.0
  Mild | 70.0
  Moderate | 10.0
  Severe | 0.0

27. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Total Aortic Regurgitation (Transvalvular & Paravalvular) (Total AR)
Time Frame: 24 months
Measure: Number; unit: percentage of participants analyzed
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 18
percentage of participants analyzed
  None | 11.1
  Trace | 38.9
  Mild | 44.4
  Moderate | 5.6
  Severe | 0.0

28. Secondary Outcome: Repeat Hospitalization
Time Frame: 0 day to 30 days
Measure: Number; unit: prob of freedom from event @ 30 days
Arm/Group | As Treated Subjects
Number analyzed (Participants) | 20
prob of freedom from event @ 30 days | 80.0

29. Secondary Outcome: Repeat Hospitalization
Time Frame: 0 day to 6 months
Measure: Number; unit: prob of freedom from event @ 183 days
Arm/Group | As Treated Subjects
Number analyzed (Participants) | 20
prob of freedom from event @ 183 days | 55.0

30. Secondary Outcome: Repeat Hospitalization
Time Frame: 0 day to 12 months
Measure: Number; unit: prob of freedom from event @ 365 days
Arm/Group | As Treated Subjects
Number analyzed (Participants) | 20
prob of freedom from event @ 365 days | 35.0

31. Secondary Outcome: Repeat Hospitalization
Time Frame: 0 day to 24 months
Measure: Number; unit: prob of freedom from event @ 730 days
Arm/Group | As Treated Subjects
Number analyzed (Participants) | 20
prob of freedom from event @ 730 days | 30.0

32. Secondary Outcome: Valve-related Deaths
Time Frame: 0 day to 30 days
Measure: Number; unit: prob of freedom from event @ 30 days
Arm/Group | As Treated Subjects
Number analyzed (Participants) | 20
prob of freedom from event @ 30 days | 100.0

33. Secondary Outcome: Valve-related Deaths
Time Frame: 0 day to 6 months
Measure: Number; unit: prob of freedom from event @ 183 days
Arm/Group | As Treated Subjects
Number analyzed (Participants) | 20
prob of freedom from event @ 183 days | 100.0

34. Secondary Outcome: Valve-related Deaths
Time Frame: 0 day to 12 months
Measure: Number; unit: prob of freedom from event @ 365 days
Arm/Group | As Treated Subjects
Number analyzed (Participants) | 20
prob of freedom from event @ 365 days | 100.0

35. Secondary Outcome: Valve-related Deaths
Time Frame: 0 day to 24 months
Measure: Number; unit: prob of freedom from event @ 730 days
Arm/Group | As Treated Subjects
Number analyzed (Participants) | 20
prob of freedom from event @ 730 days | 100

36. Secondary Outcome: Quality of Life Assessment Using SF-36 Questionnaire - Physical Component Summary (Paired Change From Baseline)
Description: The SF-36 assessment was used to evaluate subject Quality of life (QoL) by assessing change in physical function and general health status. The SF-36 v2 ͭ ͫ Scoring Program was used to convert raw scores ranging from 0 to 100 into norm-based scores, allowing direct comparison to the reference values for the Japanese population. The Z-score of each subdomain is calculated as the numbers of standard deviation away from the Japanese population mean of the corresponding raw score. Norm-based score is then derived as fifty plus 10 times of the z-score. A norm-based score of less than 50 was interpreted as below average when compared to the Japanese population whereas norm-based scores greater than 50 were interpreted as above average.
Time Frame: Baseline to 30 days
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
points | 5.1 [-12.2 to 18.0]

37. Secondary Outcome: Quality of Life Assessment Using SF-36 Questionnaire - Physical Component Summary (Paired Change From Baseline)
Description: as for outcome 36
Time Frame: Baseline to 6 months
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
points | 1.7 [-12.6 to 16.3]

38. Secondary Outcome: Quality of Life Assessment Using SF-36 Questionnaire - Physical Component Summary (Paired Change From Baseline)
Description: as for outcome 36
Time Frame: Baseline to 12 months
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 20
points | 4.6 [-9.5 to 15.7]

39. Secondary Outcome: Quality of Life Assessment Using SF-36 Questionnaire - Physical Component Summary (Paired Change From Baseline)
Description: as for outcome 36
Time Frame: Baseline to 24 months
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 18
points | 5.3 [-8.0 to 19.8]

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) must be reported to the study sponsor by the investigator or study staff within 24 hours after the investigator first learns of event.
Groups:
- Iliofemoral (As Treated Subjects): The iliofemoral approach is used as the primary access site because there is a large body of clinical data in the past using this approach in patients implanted with Transcatheter Aortic Valve Implantation (TAVI) using the 23 mm MDT-2111 system.
- Direct Aortic (As Treated Subjects): For patients who would benefit from the therapy but have unfavorable non-aortic vasculature of the transfemoral and subclavian/axillary access sites (i.e. excessive atherosclerosis, calcifications, or tortuosity of arteries), the direct aortic approach is currently being used in overseas (EU and US) in clinical practice with similar outcomes to transfemoral and subclavian/ axillary artery approaches with the Transcatheter Aortic Valve Implantation (TAVI) using the 23 mm MDT-2111 system.
- All Subjects (As Treated Subjects): This includes subjects from all access approaches, iliofemoral and direct aortic who were implanted with the Transcatheter Aortic Valve Implantation (TAVI) using the 23 mm MDT-2111 system.
Arm/Group | Iliofemoral (As Treated Subjects) | Direct Aortic (As Treated Subjects) | All Subjects (As Treated Subjects)
Serious Adverse Events (participants affected / at risk) | 13/16 | 3/4 | 16/20
Other Adverse Events (participants affected / at risk) | 16/16 | 4/4 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iliofemoral (As Treated Subjects) (N=16) | Direct Aortic (As Treated Subjects) (N=4) | All Subjects (As Treated Subjects) (N=20)
Aortic Valvular Disorders (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac Conduction Disorders (Cardiac disorders) | 4 (4) | 0 (0) | 4 (4)
Cardiac Disorders Nec (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Heart Failures Nec (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Pericardial Disorders Nec (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Supraventricular Arrhythmias (Cardiac disorders) | 2 (3) | 0 (0) | 2 (3)
Blindness (Excl Colour Blindness) (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Cataract Conditions (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Non-Site Specific Gastrointestinal Haemorrhages (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oesophageal Stenosis And Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Device Issues Nec (General disorders) | 1 (1) | 1 (1) | 2 (2)
Hepatic Fibrosis And Cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatocellular Damage And Hepatitis Nec (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac Infections (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Influenza Viral Infections (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lower Respiratory Tract And Lung Infections (Infections and infestations) | 4 (4) | 0 (0) | 4 (4)
Sepsis, Bacteraemia, Viraemia And Fungaemia Nec (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal Infections (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Lower Limb Fractures And Dislocations (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Skull Fractures, Facial Bone Fractures And Dislocations (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Spinal Fractures And Dislocations (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Total Fluid Volume Decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Arthropathies Nec (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Breast And Nipple Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Central Nervous System Haemorrhages And Cerebrovascular Accidents (Nervous system disorders) | 0 (0) | 1 (2) | 1 (2)
Breathing Abnormalities (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax And Pleural Effusions Nec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Aortic Necrosis And Vascular Insufficiency (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Lymphangiopathies (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Non-Site Specific Necrosis And Vascular Insufficiency Nec (Vascular disorders) | 0 (0) | 1 (4) | 1 (4)
Peripheral Embolism And Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iliofemoral (As Treated Subjects) (N=16) | Direct Aortic (As Treated Subjects) (N=4) | All Subjects (As Treated Subjects) (N=20)
Anaemia Deficiencies (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Anaemias Nec (Blood and lymphatic system disorders) | 6 (7) | 2 (2) | 8 (9)
Lymphatic System Disorders Nec (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac Conduction Disorders (Cardiac disorders) | 9 (10) | 3 (4) | 12 (14)
Heart Failures Nec (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Rate And Rhythm Disorders Nec (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Supraventricular Arrhythmias (Cardiac disorders) | 4 (5) | 0 (0) | 4 (5)
Ventricular Arrhythmias And Cardiac Arrest (Cardiac disorders) | 3 (3) | 0 (0) | 3 (3)
Diarrhoea (Excl Infective) (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)
Gastrointestinal And Abdominal Pains (Excl Oral And Throat) (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Gastrointestinal Atonic And Hypomotility Disorders Nec (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4)
Nausea And Vomiting Symptoms (Gastrointestinal disorders) | 3 (3) | 2 (2) | 5 (5)
Administration Site Reactions Nec (General disorders) | 1 (1) | 1 (1) | 2 (2)
Complications Associated With Device Nec (General disorders) | 1 (1) | 0 (0) | 1 (1)
Device Physical Property And Chemical Issues (General disorders) | 1 (2) | 0 (0) | 1 (2)
Febrile Disorders (General disorders) | 1 (1) | 0 (0) | 1 (1)
Implant And Catheter Site Reactions (General disorders) | 3 (3) | 0 (0) | 3 (3)
Inflammations (General disorders) | 2 (2) | 0 (0) | 2 (2)
Infusion Site Reactions (General disorders) | 1 (1) | 0 (0) | 1 (1)
Oedema Nec (General disorders) | 1 (1) | 2 (2) | 3 (3)
Pain And Discomfort Nec (General disorders) | 1 (1) | 1 (2) | 2 (3)
Hepatic And Hepatobiliary Disorders Nec (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Hepatic Enzymes And Function Abnormalities (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Herpes Viral Infections (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Infections Nec (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Influenza Viral Infections (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Upper Respiratory Tract Infections (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary Tract Infections (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Fractures And Dislocations Nec (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Non-Site Specific Injuries Nec (Injury, poisoning and procedural complications) | 4 (6) | 1 (2) | 5 (8)
Non-Site Specific Procedural Complications (Injury, poisoning and procedural complications) | 1 (2) | 2 (3) | 3 (5)
Skin Injuries Nec (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Spinal Fractures And Dislocations (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Carbohydrate Tolerance Analyses (Incl Diabetes) (Investigations) | 1 (1) | 0 (0) | 1 (1)
Liver Function Analyses (Investigations) | 6 (6) | 2 (2) | 8 (8)
Metabolism Tests Nec (Investigations) | 6 (6) | 2 (2) | 8 (8)
Mineral And Electrolyte Analyses (Investigations) | 1 (1) | 1 (1) | 2 (2)
Platelet Analyses (Investigations) | 7 (7) | 3 (4) | 10 (11)
Protein Analyses Nec (Investigations) | 9 (11) | 3 (4) | 12 (15)
Renal Function Analyses (Investigations) | 1 (1) | 1 (1) | 2 (2)
Skeletal And Cardiac Muscle Analyses (Investigations) | 4 (4) | 2 (3) | 6 (7)
Tissue Enzyme Analyses Nec (Investigations) | 3 (3) | 1 (1) | 4 (4)
Vascular Tests Nec (Incl Blood Pressure) (Investigations) | 4 (5) | 1 (2) | 5 (7)
White Blood Cell Analyses (Investigations) | 1 (1) | 1 (1) | 2 (2)
Hyperlipidaemias Nec (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Lipid Metabolism And Deposit Disorders Nec (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Potassium Imbalance (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 4 (4)
Protein Metabolism Disorders Nec (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 4 (4)
Joint Related Signs And Symptoms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Muscle Related Signs And Symptoms Nec (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal And Connective Tissue Pain And Discomfort (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 5 (6)
Musculoskeletal And Connective Tissue Signs And Symptoms Nec (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Rheumatoid Arthropathies (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Soft Tissue Disorders Nec (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Central Nervous System Haemorrhages And Cerebrovascular Accidents (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Headaches Nec (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Memory Loss (Excl Dementia) (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Neurological Signs And Symptoms Nec (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Structural Brain Disorders Nec (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Confusion And Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Disturbances In Initiating And Maintaining Sleep (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (2)
Urinary Abnormalities (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Breathing Abnormalities (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Coughing And Associated Symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Lower Respiratory Tract Inflammatory And Immunologic Conditions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nasal Disorders Nec (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3)
Pneumothorax And Pleural Effusions Nec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis Ascribed To Specific Agent (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rashes, Eruptions And Exanthems Nec (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Skin Haemorrhages (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 4 (4)
Blood Pressure Disorders Nec (Vascular disorders) | 0 (0) | 2 (2) | 2 (2)
Haemorrhages Nec (Vascular disorders) | 2 (2) | 0 (0) | 2 (2)
Lymphangiopathies (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Lymphoedemas (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral Aneurysms And Dissections (Vascular disorders) | 3 (3) | 0 (0) | 3 (3)
Vascular Hypotensive Disorders (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No